CLINICAL TRIAL: NCT01364922
Title: A Phase 2, Randomized Withdrawal Study of the Analgesic Efficacy and Safety of Hydrocodone/Acetaminophen Extended Release Compared to Placebo in Subjects With Chronic Low Back Pain
Brief Title: Phase 2 Chronic Low Back Pain Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-807
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open-label Hydrocodone/Acetaminophen Extended Release (Experimental): Hydrocodone/acetaminophen extended release, 2 tablets twice daily
  Interventions: Drug: hydrocodone/acetaminophen extended release
- Double-blind Hydrocodone/Acetaminophen Extended Release (Experimental): Hydrocodone/acetaminophen extended release, 1 tablet twice daily
  Interventions: Drug: hydrocodone/acetaminophen extended release
- Double-blind Placebo (Placebo Comparator): Placebo, 1 tablet twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydrocodone/acetaminophen extended release
  Other Names: ABT-712
  Arms: Double-blind Hydrocodone/Acetaminophen Extended Release; Open-label Hydrocodone/Acetaminophen Extended Release
Drug: Placebo
  Arms: Double-blind Placebo

SUMMARY:
The primary purpose of this study was to evaluate the analgesic effect and safety of hydrocodone/acetaminophen extended release compared to placebo.

DETAILED DESCRIPTION:
This phase 2, multicenter, double-blind (DB), placebo-controlled, randomized withdrawal study compared the analgesic efficacy and safety of hydrocodone/acetaminophen extended release to placebo in subjects with moderate to moderately severe chronic lower back pain (CLBP). Participants met pre-defined criteria at the conclusion of the open-label (OL) Titration Period to proceed to randomization into the double-blind (DB) Maintenance Period of the study. Study drug was given for a total of approximately 5 weeks, which included 2 weeks in OL, 2 weeks in DB, and a 3-day taper. During the OL period, all participants took increasing doses of hydrocodone/acetaminophen extended release until they were taking 2 tablets, twice daily. During the DB period, participants in the hydrocodone/acetaminophen extended release group took 1 hydrocodone/acetaminophen extended release tablet twice daily throughout the 2 weeks, while participants in the placebo group took 1 placebo tablet twice daily.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects who have a diagnosis of chronic low back pain of at least 6 month duration

Exclusion Criteria:

Subjects with a history of surgical or invasive intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Quintana Diez, MD, Study Director — AbbVie
Locations (17):
- United States (17):
  - Site Reference ID/Investigator# 54875, Tucson, Arizona
  - Site Reference ID/Investigator# 54876, Anaheim, California
  - Site Reference ID/Investigator# 54877, Burbank, California
  - Site Reference ID/Investigator# 54873, Lomita, California
  - Site Reference ID/Investigator# 54874, DeLand, Florida
  - Site Reference ID/Investigator# 54866, Oldsmar, Florida
  - Site Reference ID/Investigator# 54879, Marietta, Georgia
  - Site Reference ID/Investigator# 54865, Valparaiso, Indiana
  - Site Reference ID/Investigator# 54782, Prairie Village, Kansas
  - Site Reference ID/Investigator# 54862, Pasadena, Maryland
  - Site Reference ID/Investigator# 54878, Watertown, Massachusetts
  - Site Reference ID/Investigator# 54880, St Louis, Missouri
  - Site Reference ID/Investigator# 54881, Williamsville, New York
  - Site Reference ID/Investigator# 54872, Cincinnati, Ohio
  - Site Reference ID/Investigator# 54863, Marion, Ohio
  - Site Reference ID/Investigator# 54745, Killeen, Texas
  - Site Reference ID/Investigator# 54742, San Antonio, Texas

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Hydrocodone/Acetaminophen Extended Release: 2 hydrocodone/acetaminophen extended release tablets, twice daily, for 2 weeks.
- Double-blind Hydrocodone/Acetaminophen Extended Release: 1 hydrocodone/acetaminophen extended release tablet, twice daily, for 2 weeks.
- Double-blind Placebo: 1 placebo tablet, twice daily, for 2 weeks.
Period: Open-label (OL) Period
Arm/Group | Open-label Hydrocodone/Acetaminophen Extended Release | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Started | 168 | 0 | 0
Completed | 146 | 0 | 0
Not Completed | 22 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Did Not Meet Randomization Criteria | 6 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other, Unspecified | 1 | 0 | 0
Period: Double-Blind (DB) Period
Arm/Group | Open-label Hydrocodone/Acetaminophen Extended Release | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Started | 0 | 99 | 47
Completed | 0 | 94 | 42
Not Completed | 0 | 5 | 5
Not completed — Lack of Efficacy | 0 | 3 | 4
Not completed — Subject Noncompliant | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Other, Unspecified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OL Hydrocodone/Acetaminophen Extended Release (Nonrandomized): 2 hydrocodone/acetaminophen extended release tablets, twice daily, for 2 weeks. These participants enrolled in the study and received at least one dose of study drug during the open-label period; these participants were not randomized and did not progress to the double-blind period.
- DB Hydrocodone/Acetaminophen Extended Release: 1 hydrocodone/acetaminophen extended release tablet, twice daily, for 2 weeks. These participants completed the open-label period (hydrocodone/acetaminophen extended release, 2 tablets twice daily), and were randomized to receive hydrocodone/acetaminophen extended release during the double-blind period.
- DB Placebo: 1 placebo tablet, twice daily, for 2 weeks. These participants completed the open-label period (hydrocodone/acetaminophen extended release, 2 tablets twice daily), and were randomized to receive placebo during the double-blind period.
- Total: Total of all reporting groups
Arm/Group | OL Hydrocodone/Acetaminophen Extended Release (Nonrandomized) | DB Hydrocodone/Acetaminophen Extended Release | DB Placebo | Total
Number analyzed (Participants) | 22 | 99 | 47 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.82) | 47.9 (13.62) | 52.7 (13.82) | 49.7 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 61 | 30 | 106
  Male | 7 | 38 | 17 | 62
Double-blind Baseline Chronic Lower Back Pain (CLBP) Intensity VAS [Mean (Standard Deviation); unit: scores on a scale] — The last assessment using the CLBP Intensity Visual Analog Scale (VAS) (0 mm = No Pain and 100 mm = Worst Pain Imaginable) conducted before the first dose in the double blind period.
  scores on a scale | NA (NA) — These subjects were not randomized to the double-blind period. | 26.9 (13.78) | 31.7 (11.17) | 28.5 (13.14)
Double-blind Participant's Global Assessment of Back Pain Status [Number; unit: participants] — Participant answered the question "Considering all the ways your chronic low back pain affects you, how are you doing today?" on a 5-point scale: very good (no symptoms and no limitation of normal activities); good (mild symptoms and no limitation of normal activities); fair (moderate symptoms and limitation of some normal activities); poor (severe symptoms and inability to carry out most normal activities); very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Values presented for all participants with double-blind baseline data.
  participants
    Fair | NA — These subjects were not randomized to the double-blind period. | 21 | 14 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Good | NA — These subjects were not randomized to the double-blind period. | 57 | 29 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Poor | NA — These subjects were not randomized to the double-blind period. | 2 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Very Good | NA — These subjects were not randomized to the double-blind period. | 15 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Change From Double-blind Baseline in Chronic Lower Back Pain (CLBP) Intensity by Visual Analog Scale (VAS)
Description: The change from the double-blind randomization baseline (DB baseline: the last assessment before first dose in the double-blind period) to the final assessment in pain intensity, assessed using the CLBP Intensity VAS (0 mm = No Pain and 100 mm = Worst Pain Imaginable). Least squares means and standard errors from an ANCOVA model.
Time Frame: Double-blind baseline to Day 29
Population: The analysis of the primary outcome measure included all randomized participants who received at least 1 dose of study drug during the double-blind period (double-blind intent-to-treat) and had at least 1 assessment during the double-blind period.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Number analyzed (Participants) | 95 | 46
scores on a scale | 10.9 (2.86) | 19.9 (3.77)

2. Secondary Outcome: Participant's Global Assessment of Back Pain Status at Final Evaluation
Description: The participant's overall impression of their back pain status was obtained by having the participant answer the question "Considering all the ways your chronic low back pain affects you, how are you doing today?" on a 5-point categorical scale: very good (no symptoms and no limitation of normal activities); good (mild symptoms and no limitation of normal activities); fair (moderate symptoms and limitation of some normal activities); poor (severe symptoms and inability to carry out most normal activities); very poor (very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Double-blind baseline to Day 29
Measure: Number; unit: participants
Arm/Group | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Number analyzed (Participants) | 95 | 46
participants
  Very Good | 13 | 2
  Good | 47 | 16
  Fair | 25 | 19
  Poor | 10 | 9
  Very Poor | 0 | 0

3. Secondary Outcome: Participant's Global Assessment of Study Drug at Final Evaluation
Description: The participant's overall impression of the study drug was obtained by having the participant answer the question "How would you rate your overall response to the study medication?" on a 5-point categorical scale: excellent; very good; good; fair; poor.
Time Frame: Double-blind baseline to Day 29
Population: Double-blind intent to treat population; scores for participants with no post-randomization assessment were excluded from this analysis.
Measure: Number; unit: participants
Arm/Group | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Number analyzed (Participants) | 93 | 46
participants
  Excellent | 2 | 7
  Very Good | 11 | 4
  Good | 36 | 19
  Fair | 31 | 11
  Poor | 13 | 5

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time of study drug administration to 30 days after last dose (total 9 weeks); SAEs were recorded from the time that informed consent was obtained until 30 days following discontinuation of study drug (total 13 weeks).
Description: AEs with onset during the OL period are shown separately from AEs with onset after the first dose of study drug (hydrocodone/acetaminophen extended release or placebo) in the DB period.
Groups:
- Open-label Hydrocodone/Acetaminophen Extended Release: 2 hydrocodone/acetaminophen extended release tablets, twice daily, for 2 weeks. These participants enrolled in the study and received at least one dose of study drug during the open-label period.
- Double-blind Hydrocodone/Acetaminophen Extended Release: 1 hydrocodone/acetaminophen extended release tablet, twice daily, for 2 weeks. These participants completed the open-label period (hydrocodone/acetaminophen extended release, 2 tablets twice daily), and were randomized to receive hydrocodone/acetaminophen extended release during the double-blind period.
- Double-blind Placebo: 1 placebo tablet, twice daily, for 2 weeks. These participants completed the open-label period (hydrocodone/acetaminophen extended release, 2 tablets twice daily), and were randomized to receive placebo during the double-blind period.
Arm/Group | Open-label Hydrocodone/Acetaminophen Extended Release | Double-blind Hydrocodone/Acetaminophen Extended Release | Double-blind Placebo
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/99 | 1/47
Other Adverse Events (participants affected / at risk) | 70/168 | 7/99 | 8/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Hydrocodone/Acetaminophen Extended Release (N=168) | Double-blind Hydrocodone/Acetaminophen Extended Release (N=99) | Double-blind Placebo (N=47)
CHEST PAIN (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Hydrocodone/Acetaminophen Extended Release (N=168) | Double-blind Hydrocodone/Acetaminophen Extended Release (N=99) | Double-blind Placebo (N=47)
CONSTIPATION (Gastrointestinal disorders) | 32 | 3 | 2
NAUSEA (Gastrointestinal disorders) | 22 | 2 | 4
DIZZINESS (Nervous system disorders) | 18 | 0 | 1
HEADACHE (Nervous system disorders) | 9 | 1 | 3
SOMNOLENCE (Nervous system disorders) | 13 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.